CLINICAL TRIAL: NCT06824129
Title: Clinical Performance Evaluation of the QIAstat-Dx® cUTI Plus AMR Panel on Patients Suspected of Complicated Urinary Tract Infection
Brief Title: Clinical Performance Evaluation of the QIAstat-Dx® cUTI Plus AMR
Status: Active, not recruiting | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF-19-0598-0-CSP-001
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Complicated Urinary Tract Infection
Keywords: QIAstat-Dx; Clinical Performance Study; complicated Urinary infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Performance evaluation of QIAstat-Dx cUTI Plus AMR Panel using the QIAstat-Dx® Analyzer to demonstrate that the QIAstat-Dx cUTI Plus AMR Panel achieves its intended performance during normal conditions of use by the intended user in the intended environment

DETAILED DESCRIPTION:
The objective of the study is to demonstrate that the QIAstat-Dx cUTI Plus AMR Panel achieves its intended performance during normal conditions of use by the intended user in the intended environment.

The primary objective is to evaluate the performance of QIAstat-Dx cUTI Plus AMR Panel in comparison with the results obtained from the reference method.

The secondary objective of the study is to evaluate the safety ofQIAstat-Dx cUTI Plus AMR Panel with respect to users/operators.

The primary study endpoint will be the results for each analyte obtained from testing prospective specimens with QIAstat-Dx cUTI Plus AMR Panel and Reference Method. Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) will be determined

ELIGIBILITY:
Inclusion Criteria:

* Specimens from subjects of all ages and demographic characteristics can be enrolled.

  * Specimen must come from patients with suspected cUTI by their healthcare provider:
  * Urine specimen with evidence of pyuria confirmed by positive urine analysis (Dipstick analysis positive for leukocyte esterase or at least 10 White Blood Cells percubic millimeter) And
  * A sign or symptom of a cUTI (for example: chills or rigors or warmth associated with fever, malaise, flank pain or pelvic pain and/or costo-vertebral angle pain or tenderness on physical examination, nausea or vomiting, dysuria, urinary frequency or urinary urgency)
  * Specimen must be residual leftover and de-identified
  * Specimen obtained preserved (containing boric acid, sodium formate or sodium borate) or unpreserved as midstream urine or fresh urine catheter
  * For Preserved Only: Fresh prospectively collected preserved specimens stored to up 48 hours at 15°C-25°C or 24 hours at 2°C-8°C.
  * For Unpreserved Only: Fresh prospectively collected unpreserved specimens stored up to 24 hours at 2°C-8°C.
  * Specimen must have a minimum of 3 ml of urine available.
  * Specimen date of collection and standard of Care testing results should be available.
  * Specimen must be unique (only one sample enrolled per patient).

Exclusion Criteria:

* Specimens enrolled in the study may be excluded for the following reasons:

  * Lack of clear subject identification or label on urine specimen.
  * Specimen has been centrifuged.
  * Obvious physical damage of residual specimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with signs and symptoms of complicated urine infection
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
PPA | 8 months
  Positive percent agreement
NPA | 8 months
  Negative percent agreement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Principal Investigator — Qiagen Manchester Limited
Locations (1):
- QIAGEN, Manchester, United Kingdom